CLINICAL TRIAL: NCT04744428
Title: Test of an Innovative, Scalable Support Program for Parents With a Young Child Recently Diagnosed With Autism Spectrum Disorder
Brief Title: Trial of Autism Parent Navigator Program
Acronym: APN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of South Carolina (Other); Family Connections (Unknown)
Responsible Party: Principal Investigator, Mark Feinberg, Research Professor, Feinberg, Mark, Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: APN-RT01
Record Dates: First submitted 2020-04-09; First posted 2021-02-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Parent Navigators Intervention (Experimental): Autism Parent Navigators Intervention is a manualized, in-home, peer support model for parents with a young child recently diagnosed with ASD.
  Interventions: Behavioral: Autism Parent Navigators
- Peer mentoring (Active Comparator): Peer mentors will offer an equivalent number of in-home or telephone visits for families, providing non-manualized peer support.
  Interventions: Behavioral: Peer mentoring

INTERVENTIONS:
Behavioral: Autism Parent Navigators — The Autism Parent Navigator program consists of six sessions delivered to parents in the home, supporting adjustment to ASD, accessing services, and coparenting support.
  Arms: Autism Parent Navigators Intervention
Behavioral: Peer mentoring — Six in-home or telephone sessions, depending on family uptake, providing non-manualized general support as usual from parent peer mentors regarding adjustment to ASD.
  Arms: Peer mentoring

SUMMARY:
To address the dual needs of parents for support in navigating Autistic Spectrum Disorder (ASD) services and maintaining positive family functioning, the investigators propose to test Autism Parent Navigators (APN), an innovative in-home, peer support model for parents with a young child recently diagnosed with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children who have been newly diagnosed with Autism Spectrum Disorder (ASD).
* The child will be age 2-6 years and been diagnosed with ASD in the past four months.
* The child is the first child in the family to be diagnosed with ASD.
* Parents are not already involved in a parent mentoring relationship.
* Parents are currently involved in a couple relationship, including same-sex partners, dating couples, adoptive parents and step-parent families.

Exclusion Criteria:

None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Weekly Count of Service Navigation Behaviors | 12 month
  Engagement with ASD-related Services
Parenting Scale (Arnold) | 12 month
  Parenting consistency, warmth
CES-Depression | 12 month
  Parent depression

SECONDARY OUTCOMES:
Coparenting Relationship Scale (Feinberg, Brown, & Kan, 2012) | 12 month
  Coparenting Support
Family Empowerment Scale - FES | 12 month
  Parent Efficacy regarding Service Access
PDD-BI | 12 month
  Challenging Child Behaviors: Aggression, Non-compliance

CONTACTS AND LOCATIONS:
Overall Officials: Mark Feinberg, PhD, Principal Investigator — Penn State
Locations (1):
- USC, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No